CLINICAL TRIAL: NCT02958202
Title: A Multi Center, Multi National, Open Label, Extension Study to Evaluate the Long-term Efficacy and Safety of BMN 044 (PRO044) in Subjects With Duchenne Muscular Dystrophy
Brief Title: Extension Study of BMN 044 in Duchenne Muscular Dystrophy (DMD)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Regulatory approval was not obtained for drisapersen, hence BioMarin is stopping the development of all exon skipping oligonucleotides in DMD.
Sponsor: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BMN-044-201; 2015-003681-87 (EudraCT Number)
Record Dates: First submitted 2016-10-27; First posted 2016-11-08 (Estimated); Last update posted 2018-01-26 (Actual); Status verified 2018-01

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Duchenne Muscular Dystrophy; DMD; Dystrophin; BMN 044; PRO044; BioMarin
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- BMN 044 IV 6 mg/kg (Experimental): Weekly intravenous (IV) dosing with 6 mg/kg
  Interventions: Drug: BMN 044 IV 6 mg/kg
- BMN 044 IV 9 mg/kg (Experimental): Weekly intravenous (IV) dosing with 9 mg/kg
  Interventions: Drug: BMN 044 IV 9 mg/kg
- BMN 044 SC 6 mg/kg (Experimental): Weekly subcutaneous (SC) dosing with 6 mg/kg
  Interventions: Drug: BMN 044 SC 6 mg/kg

INTERVENTIONS:
Drug: BMN 044 IV 6 mg/kg
  Other Names: PRO044
  Arms: BMN 044 IV 6 mg/kg
Drug: BMN 044 IV 9 mg/kg
  Other Names: PRO044
  Arms: BMN 044 IV 9 mg/kg
Drug: BMN 044 SC 6 mg/kg
  Other Names: PRO044
  Arms: BMN 044 SC 6 mg/kg

SUMMARY:
The aim of this study is to provide continuing access to BMN 044 treatment for subjects previously treated with BMN 044. The information gained from this study is expected to further characterize the efficacy and safety of BMN 044 over a longer treatment period.

DETAILED DESCRIPTION:
This is a phase 2 multi center, multi national, open label, long term extension study. Up to approximately 50 male subjects with Duchenne Muscular Dystrophy (DMD) who have previously been treated with BMN 044 will be enrolled. Subjects will receive either IV infusions or SC injections at pre-defined doses.

Safety and tolerability, pharmacokinetics (PK), pharmacodynamics (PD) and efficacy assessments will be conducted at regular intervals throughout the study.

Subjects will be permitted to continue in this study until the subject meets any of the defined withdrawal criteria, BioMarin decides to halt the clinical development of BMN 044, or BMN 044 receives marketing authorization.

ELIGIBILITY:
Inclusion Criteria:

* Subjects previously treated with BMN 044 or a comparator treatment in a BMN 044 Sponsored Study or Investigator Initiated Trial and who are not eligible for another ongoing BMN 044 study.
* Continued use of glucocorticosteroids for a minimum of 60 days prior to study entry with a reasonable expectation that the subject will remain on glucocorticosteroids for the duration of this study.
* Willing and able to comply with all study requirements and procedures.
* Willing and able to provide written, signed informed consent, or in the case of subjects under the age of 18 years(or 16 years, depending on the region), provide written assent (if required) and written informed consent by a legally authorized representative after the nature of the study has been explained, and prior to the conduct of any research-related procedures.

Exclusion Criteria:

* Subjects who have previously been treated with BMN 044 who had a serious adverse experience or met safety stopping criteria, that remains unresolved, which in the opinion of the Investigator could have been attributable to BMN 044.
* History of significant medical disorder which may confound the interpretation of safety data
* Acute illness within 4 weeks prior to the first dose of BMN 044 (Week 1) which may interfere with the measurements.
* Symptomatic cardiomyopathy.
* Baseline aPTT above the upper limit of normal (ULN).
* Baseline platelet count below the lower limit of normal (LLN).
* Use of anti coagulants, anti thrombotics or anti platelet agents within 28 days of the baseline visit.
* Prior use of any investigational product (other than BMN 044) or investigational medical device must be discussed with the Medical Monitor prior to screening.
* Current or history of drug and/or alcohol abuse.

Min Age: 5 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2016-04; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Number of subjects with 1 or more treatment emergent adverse events following BMN044 dosing | Through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Paulatsya Joshi, Study Director — BioMarin Pharmaceutical
Locations (5):
- Universitair Ziekenhuis Leuven, Leuven, Belgium
- Italy (2):
  - S.Anna Hospital, Ferrara
  - Policlinico Univsersitario Agostino Gemelli, Rome
- Leiden University Medical Center, Leiden, Netherlands
- Drottning Silvias Barn- ochungdomssjukhus, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No